CLINICAL TRIAL: NCT01661608
Title: Gastric Restriction Using the EndoSurgical Operating System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA indicated study should have had prior IDE submission & approval
Sponsor: USGI Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TPR41122
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: Gastric Restriction
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EOS (Experimental): Collecting data on the use of the EOS for gastric tissue approximation during primary gastric restrictive procedures
  Interventions: Device: Using the EOS for gastric restriction

INTERVENTIONS:
Device: Using the EOS for gastric restriction

SUMMARY:
The primary objective is to collect data on the use of the EndoSurgical Operating System (EOS) for gastric tissue approximation during primary gastric restrictive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient has met diabetic lab testing and all pre-procedural qualifications as delineated below.
* Patient is >/= 20 yrs. of age and </= 60 yrs. of age
* Patient has a BMI of >/=30 and < 40
* Patient has history of obesity for >/= 2 yrs.
* Patient has had not significant weight change (<5% of total body weight) in last 6 months.
* Patient is a reasonable candidate for general anesthesia
* Patient agrees not to have any additional weight loss surgery or liposuction for 2 yrs. following procedure.

Exclusion Criteria:

* Patient is not able and willing to return for all follow-up evaluations, tests and nutritional counseling.
* Patient is not able to provide written informed consent
* Patient has history or present use of insulin or insulin derivatives for treatment of diabetes.
* Patient has diabetes secondary to a specific disease.
* Patient has history of inflammatory disease of GI tract
* Patient has diabetic retinopathy
* Patient has chronic pancreatic disease
* Patient ahs active peptic ulcer
* Patient has portal hypertension
* Patient has esophageal varices
* Patient has significant esophageal disease
* Patient has a history of any significant abdominal surgery
* Patient has a history of any bariatric or GERD surgical procedures
* Patient has a hiatal hernia > 2cm.
* Patient has esophageal stricture or other anatomy and/or condition that could preclude passage of endolumenal instruments
* Patient is of childbearing age and not practicing effective birth control method, pregnant or lactating.
* Patient has had a MI or CVA in last year, or has unstable cardiovascular disease.
* Patient has cancer or life expectancy of < 2 yrs.
* Patient currently uses or has used over the counter or prescription weight loss drugs in last month or intends to use during follow-up Registry period.
* Patient has quit smoking within last 6 months or plans to quit smoking in the next year.
* Patient has a history of durg or alcohol abuse
* Patient has uncontrolled depression, psychosis, or eating disorder.
* Patient is non-ambulatory or has significant impairment of mobility.
* Patient has known hormonal or genetic cause for obesity.
* Patient is participating in another Registry and/or Study that could adversely affect this Registry.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation in regards to Weight Loss | 24 Months Post-op

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Thomas, MD, FACS, Principal Investigator — SSL; Thomas Lavin, MD, Principal Investigator — SSL; David Voelinger, MD, Principal Investigator — Presbyterian; Peter Denk, MD, Principal Investigator — Bluegrass; Christopher Thompson, MD, Principal Investigator — Brigham & Womans; Santiago Horgan, MD, Principal Investigator — UCSD
Locations (5):
- United States (4):
  - Bluegrass, Lexington, Kentucky
  - SSL, New Orleans, Louisiana
  - Brigham & Womens, Boston, Massachusetts
  - Presbyterian, Charlotte, North Carolina
- Mexico, Mexico City, Mexico